CLINICAL TRIAL: NCT03858231
Title: The Effects of Combination Therapy of Opioids Versus Non-Opioids on Postoperative Pain Management After Knee Arthroscopic Surgery: A Prospective Randomized Controlled Study
Brief Title: Opioids Versus Non-Opioids Postoperative After Knee Arthroscopic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH Opioid Knee
Record Dates: First submitted 2019-02-19; First posted 2019-02-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Knee Injuries; Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Knee Injuries; Pain, Postoperative | interventions — oxycodone-acetaminophen; Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid (Active Comparator)
  Interventions: Drug: Norco 5Mg-325Mg Tablet
- Non-opioid (Active Comparator)
  Interventions: Drug: Ibuprofen 600 mg; Drug: Acetaminophen 325Mg Tab

INTERVENTIONS:
Drug: Norco 5Mg-325Mg Tablet — 1 tablet up to 4 times per day for 7 days
  Arms: Opioid
Drug: Ibuprofen 600 mg — 1 tablet up to 4 times per day for 7 days
  Arms: Non-opioid
Drug: Acetaminophen 325Mg Tab — 1 tablet up to 4 times per day for 7 days
  Arms: Non-opioid

SUMMARY:
The purpose of this study is to look at pain management with opioids versus non-opioids after knee arthroscopy. This study will determine 1) whether the most commonly used non-narcotic medications provide pain relief comparable with the most commonly prescribed narcotic medications in patients undergoing arthroscopic knee surgery, and 2) whether patients' characteristics (gender, pre-operative knee symptoms, workers compensation status and employment status) affect pain level following surgery or medication usage.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years of age through ≤ 80 years of age
2. Subjects undergoing elective arthroscopic knee surgery, to include partial meniscectomy, chondroplasty, or loose body removal.

Exclusion Criteria:

1. Previously enrolled in this study (enrolled for contralateral knee in this study)
2. Knee arthroscopy patients scheduled for knee ligament reconstructions
3. Bilateral knee arthroscopy
4. History of chronic opioid use or long-term analgesic therapy
5. Documented or suspected substance abuse
6. Documented or suspected chronic pain syndrome
7. Any known allergy or adverse reaction or contraindication to the components of hydrocodone, acetaminophen, or ibuprofen
8. History or symptoms of any significant medical problem in the last year (i.e., arrhythmia, impaired cardiovascular function, gastrointestinal bleeding, liver disease, renal disease)
9. With active peptic ulcer disease (history of severe heartburn)
10. Symptoms of infection with initial enrollment
11. Pregnant or nursing
12. Diagnosis of cognitive impairment
13. Unable or unwilling to provide informed consent for surgery or enrollment in this clinical study
14. Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by Institutional Review Board) and agree to abide by the study restrictions.
15. Patient refusal
16. Currently taking Coumadin, Plavix, anticoagulation medications, or medications that increase bleeding, with the exception of ASA 81mg.
17. Patients with other medical or psychological health conditions that preclude them from either receiving the intervention or returning for follow-up visits.
18. Alcoholism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain Assessment at 2 weeks | Daily for 2 weeks post-operatively
  Visual Analog Scale from 0 to 10 with 0 being no pain and 10 being worst possible, unbearable, excruciating pain
Change from Baseline Medication Use at 2 weeks | Daily for 14 days post-operatively
  Patients will be asked how many study medication capsules have they taken.

SECONDARY OUTCOMES:
Change from Baseline Knee Injury and Osteoarthritis Outcome Score (KOOS) at 6 weeks | baseline, 2 weeks, and 6 weeks post-operatively
  Sub-scales are listed as follows: 5 qualitative questions related to knee symptoms ranging from "never" to "always", 2 qualitative questions related to knee stiffness ranging from "none" to "extreme", 9 qualitative questions related to pain ranging from "none" to "extreme", 17 qualitative questions related to function and daily living ranging from "none" to "extreme", 5 qualitative questions related to function and sports and recreational activities ranging from "none" to "extreme", and 4 qualitative questions related to quality of life ranging from "never or not at all" to "constantly, totally, or extreme".
Change from Baseline Patient Reported Outcome Measurement Information System (PROMIS) at 6 weeks | baseline, 2 weeks, and 6 weeks post-operatively
  7 qualitative questions related to pain interference with responses ranging from "not at all" to "very much"

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Piatt, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health, Fargo, North Dakota, United States